CLINICAL TRIAL: NCT07074652
Title: The Effect of SSRIs on Threat of Shock Potentiated Neural Circuitry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCLH/UCL Joint Research Office (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 6198/002
Record Dates: First submitted 2025-06-25; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Anxiety
Keywords: anxiety; selective serotonin reuptake inhibitor; emotion; functional magnetic resonance imaging
MeSH Terms: conditions — Anxiety Disorders | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Control - Escitalopram (Active Comparator): Participants took 10mg escitalopram for 2-3 weeks, once daily. Escitalopram was administered in the form of a tablet, manufactured and donated for research by Lundbeck (tablet core: microcrystalline cellulose, colloidal anhydrous silica, croscarmellose sodium, talc, magnesium stearate; tablet coating: hypromellose 6cP, titanium dioxide (E171), macrogol 6000). Exact length of administration was dependent on participants' availability to attend their second scan.
  Interventions: Drug: Escitalopram
- Healthy Control - Placebo (Placebo Comparator): Participants took a placebo tablet for 2-3 weeks, once daily. Placebo was administered in the form of a tablet, manufactured and donated for research by Lundbeck and matching the escitalopram tablet given to the other study groups in colour and size. Exact length of administration was dependent on participants' availability to attend their second scan.
  Interventions: Drug: Placebo
- Anxious Individuals - Escitalopram (Experimental): Participants took 10mg escitalopram for 2-3 weeks, once daily. Escitalopram was administered in the form of a tablet, manufactured and donated for research by Lundbeck (tablet core: microcrystalline cellulose, colloidal anhydrous silica, croscarmellose sodium, talc, magnesium stearate; tablet coating: hypromellose 6cP, titanium dioxide (E171), macrogol 6000). Exact length of administration was dependent on participants' availability to attend their second scan.
  Interventions: Drug: Escitalopram
- Anxious Individuals - Placebo (Placebo Comparator): Participants took a placebo tablet for 2-3 weeks, once daily. Placebo was administered in the form of a tablet, manufactured and donated for research by Lundbeck and matching the escitalopram tablet given to the other study groups in colour and size. Exact length of administration was dependent on participants' availability to attend their second scan.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Participants received 2-3 weeks of escitalopram.
  Arms: Anxious Individuals - Escitalopram; Healthy Control - Escitalopram
Drug: Placebo — Participants received 2-3 weeks of placebo, matched in colour and size to the escitalopram.
  Arms: Anxious Individuals - Placebo; Healthy Control - Placebo

SUMMARY:
This study aims to increase the knowledge about psychological processes which may contribute to mental health problems such as depression and anxiety. This study aims to investigate if administering Escitalopram, an antidepressant which increases serotonin levels in parts of the brain, affects how the brain processes emotional information. It is hoped that measuring these changes will increase the understanding of processes involved in mental health problems.

ELIGIBILITY:
INCLUSION CRITERIA

Healthy Controls:

* Fluency in English
* Registration with a UK General Practitioner
* Capacity for consent
* No personal history of long-term medical conditions or psychiatric illness (including substance dependence, assessed with the Mini International Neuropsychiatric Interview)

Anxious Individuals:

* Fluency in English
* Registration with a UK General Practitioner
* Capacity for consent
* Meeting criteria for generalised anxiety disorder, panic disorder and/or agoraphobia (also assessed with the Mini International Neuropsychiatric Interview); permitted comorbid conditions were: major depressive disorder, obsessive-compulsive disorder and/or post-traumatic stress disorder

EXCLUSION CRITERIA

Healthy Controls and Anxious Individuals:

* Having consumed alcohol within 12 hours prior to the study
* having used illicit drugs within 3 months prior to the study
* Having had any contraindications to MRI scanning
* Being pregnant or breastfeeding
* Having had impaired or uncorrected vision or hearing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
'Aversive amplification circuit' connectivity | Baseline and 2-3 weeks after baseline
  The engagement of the neural circuit of the amygdala, cingulate cortex and prefrontal cortex will be measured via an fMRI analysis technique called a psychophysiological interactions (PPI) analysis. PPI analysis concerns behaviour-specific increases in the relationship across regional brain activity - this means that it can allow one to assess whether two regions (a priori selected ROIs) show increased connectivity during a specific context or behaviour, suggesting a behaviour-specific increase in transfer of information. The output of this analysis will take form of a continuous beta weight - an index of connectivity across two brain regions (amygdala and medial prefrontal cortex), which represents the primary outcome of the study.

SECONDARY OUTCOMES:
Cognitive task performance: Loss/risk aversion task | Baseline and 2-3 weeks after baseline
  Measures how averse participants are to risk and loss in a mock gambling context
Cognitive task performance: Go/no-go task | Baseline and 2-3 weeks after baseline
  Measures approach/avoidance behaviours under threat of shock or safe conditions
Cognitive task performance: Facial emotional processing task | Baseline and 2-3 weeks after baseline
  Measures brain responses to positive, negative and neutral emotions
Cognitive task performance: Emotional face recognition task | Baseline and 2-3 weeks after baseline
  Measures brain responses during two distinct memory processes - the encoding (learning) and retrieval (remembering) of information
Cognitive task performance: Visual affective bias task | Baseline and 2-3 weeks after baseline
  Measures biases in patients' cognition towards or away from rewarding stimuli
Regional activations during neuroimaging task: Facial emotional processing task | Baseline and 2-3 weeks after baseline
  Measures brain responses to positive, negative and neutral emotions
Regional activations during neuroimaging task: Emotional face recognition task | Baseline and 2-3 weeks after baseline
  Measures brain responses during two distinct memory processes - the encoding (learning) and retrieval (remembering) of information
Regional activations during neuroimaging task: Visual affective bias task | Baseline and 2-3 weeks after baseline
  Measures biases in patients' cognition towards or away from rewarding stimuli
Clinical symptom measure: Generalised Anxiety Disorder Scale (GAD-7) | Baseline and 2-3 weeks after baseline
  Measures symptoms of generalised anxiety, scored between 0-21 with higher scores indicating more severe symptoms
Clinical symptom measure: State Trait Anxiety Inventory (STAI) | Baseline and 2-3 weeks after baseline
  Measures state and trait anxiety symptoms, scored between 20-80 with higher scores indicating more severe symptoms
Clinical symptom measures: Patient Health Questionnaire (PHQ-9) | Baseline and 2-3 weeks after baseline
  Measures depressive symptoms, scored between 0-27 with higher scores indicating more severe symptoms
Clinical symptom measures: Beck's Depression Inventory (BDI) | Baseline and 2-3 weeks after baseline
  Measures depressive symptoms, scored between 0-63 with higher scores indicating more severe symptoms
Clinical symptom measures: Catastrophizing questionnaire | Baseline and 2-3 weeks after baseline
  Measures catastrophising, scored between 24-120 with higher scores indicating more severe symptoms
Clinical symptom measures: Daily Stress Inventory (DSI) | Baseline and 2-3 weeks after baseline
  Measures frequency and impact of daily stresses. Frequency scored between 0-58 and impact scored between 0-6, with higher scores indicating more severe stress
Clinical symptom measures: Behavioural Inhibition/Behavioural Activation Scales (BIS/BAS) | Baseline and 2-3 weeks after baseline
  Measures drive, fun-seeking, reward responsiveness and behavioural inhibition. Behavioural inhibition scored between 7-28, drive between 4-16, fun seeking between 4-16, and reward between 5-20, with higher scores indicating higher levels of those behaviours
Clinical symptom measures: Eysenck Impulsiveness Scale | Baseline and 2-3 weeks after baseline
  Measures impulsiveness, venturesomeness and empathy. Impulsivity scored between 0-19, venturesomeness between 0-16, empathy between 0-18, with higher scores indicating higher levels of those traits

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lukow PB, Lowther M, Pike AC, Yamamori Y, Chavanne AV, Gormley S, Aylward J, McCloud T, Goble T, Rodriguez-Sanchez J, Tuominen EW, Buehler SK, Kirk P, Robinson OJ. Amygdala activity after subchronic escitalopram administration in healthy volunteers: A pharmaco-functional magnetic resonance imaging study. J Psychopharmacol. 2024 Dec;38(12):1071-1082. doi: 10.1177/02698811241286773. Epub 2024 Oct 4. PMID 39364684
- [Derived] Lukow PB, Lowther M, Pike AC, Yamamori Y, Chavanne AV, Gormley S, Aylward J, Vera CE, McCloud T, Goble T, Rodriguez-Sanchez J, Tuominen EW, Buehler SK, Kirk P, Robinson OJ. Brain activation and connectivity after 2-3 weeks of escitalopram administration in anxiety disorders: A randomised trial. J Affect Disord. 2026 Feb 1;394(Pt B):120682. doi: 10.1016/j.jad.2025.120682. Epub 2025 Nov 13. PMID 41241072